CLINICAL TRIAL: NCT04401852
Title: Magnesium Sulphate for Fetal Neuroprotection in Full Term Deliveries
Brief Title: Magnesium Sulfate for Fetal Neuroprotection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 60
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Fetal Neuroprotection
MeSH Terms: interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MgSO4 group (Active Comparator): will receive a single bolus dose of 4g MgSO4 slowly intravenous over 15-20 minutes without maintenance dose
  Interventions: Drug: MgSo4
- placebo group (Placebo Comparator): will receive an equal volume of isotonic 0.9% saline over 15-20 minutes
  Interventions: Drug: Isotonic saline

INTERVENTIONS:
Drug: MgSo4 — a single bolus dose of 4g MgSO4 slowly intravenous over 15-20 minutes without maintenance dose.
  Other Names: magnesium sulfate
  Arms: MgSO4 group
Drug: Isotonic saline — equal volume of isotonic 0.9% saline over 15-20 minutes
  Arms: placebo group

SUMMARY:
Pregnant women diagnosed to have intrapartum fetal distress (Non reassuring or pathological changes according to NICE guidelines 2017) in any of the groups will receive the allocated treatment at least 20 minute before the procedure (emergency CS).

measures to reduce the effect of hypoxia will be applied to all participate through:

* The position of the mother will be changed to left lateral position (allow increased blood supply).
* I.V. fluid bolus (to avoid maternal dehydration).
* Oxytocin or cervical ripening agent will be discontinued.
* Fetal heart rate monitoring with cardiotocography will be attempted.
* If umbilical cord prolapse is noted, elevate the presenting fetal part until preparing for emergency operative delivery.
* After birth, Apgar score will be used to identify distress newborns that need resuscitation.

The study comprised 200 pregnant women. They were divided into two groups each are 100:

* Group A: pregnant women diagnosed to have intrapartum fetal distress who will receive MgSO4.
* Group B: pregnant women diagnosed to have intrapartum fetal distress who will receive placebo

DETAILED DESCRIPTION:
Pregnant women diagnosed to have intrapartum fetal distress (Non reassuring or pathological changes according to NICE guidelines 2017) in any of the groups will receive the allocated treatment at least 20 minute before the procedure (emergency CS).

measures to reduce the effect of hypoxia will be applied to all participate through:

* The position of the mother will be changed to left lateral position (allow increased blood supply).
* I.V. fluid bolus (to avoid maternal dehydration).
* Oxytocin or cervical ripening agent will be discontinued.
* Fetal heart rate monitoring with cardiotocography will be attempted.
* If umbilical cord prolapse is noted, elevate the presenting fetal part until preparing for emergency operative delivery.
* After birth, Apgar score will be used to identify distress newborns that need resuscitation.

The study comprised 200 pregnant women. They were divided into two groups each are 100:

* Group A: pregnant women diagnosed to have intrapartum fetal distress who will receive MgSO4.
* Group B: pregnant women diagnosed to have intrapartum fetal distress who will receive placebo

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 37 week of gestation.
* Not more than 35 years old.
* Fetal distress (perinatal asphyxia) diagnosed by CTG changes (Non reassuring or pathological changes according to NICE guidelines 2017).
* Clinical chorioamnionitis.
* Prolonged rupture of membranes

Exclusion Criteria:

* Medical disorders such as chronic hypertension, preeclampsia, eclampsia, DM, pulmonary hypertension, hepatic coma with risk of renal failure, and any renal, cardiac or pulmonary disease.
* RH -ve.
* Consanguinity.
* Preterm labor.
* Fetal malpresentation.
* Contraindications to the use of Magnesium Sulphate.
* Any indication for magnesium Sulphate therapy (seizure prophylaxis or tocolysis).
* Myasthenia gravis.
* Congenital fetal anomalies.
* Fetal growth restriction (birth weight < 10th Percentile for gestational age).
* Advanced cervical dilation (8cm).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Apgar score | 1 minute after delivery
  Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration between 0 and 10

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No